CLINICAL TRIAL: NCT04685915
Title: A Phase II Study of Copanlisib to Deepen Response in CLL Patients on Ibrutinib or Acalabrutinib in the Relapsed/Refractory Setting
Brief Title: Copanlisib Plus Ibrutinib or Acalabrutinib in R/R CLL
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Bayer is no longer funding due to lack of accrual
Sponsor: Inhye Ahn (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor-Investigator, Inhye Ahn, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-281
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2023-01

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
Keywords: Chronic Lymphocytic Leukemia (CLL); Ibrutinib; Acalabrutinib; Copanlisib
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib; copanlisib; acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Addition of copanlisib to either ibrutinib or acalabrutinib (Experimental): During the 28-day study treatment cycles, participants will:
  * Continue to take ibrutinib (daily) or acalabrutinib (twice a day) at a predetermined dose for as long as there are no serious side effects and disease progression
  * Receive intravenous infusion of copanlisib at a predetermined dose days 1, 8 and 15 for cycles 1-6.
  Interventions: Drug: Ibrutinib; Drug: Copanlisib; Drug: Acalabrutinib

INTERVENTIONS:
Drug: Ibrutinib — Capsule, taken by mouth once daily
  Other Names: Imbruvica
Drug: Copanlisib — Intravenous Infusion
  Other Names: Aliqopa
Drug: Acalabrutinib — Capsule, taken by mouth twice daily
  Other Names: Calquence

SUMMARY:
This research study is examining the effect of adding a fixed duration of copanlisib to ibrutinib or acalabrutinib in select participants who have been on ibrutinib or acalabrutinib for at least six months for relapsed/refractory chronic lymphocytic leukemia (CLL).

The names of the study drugs involved in this study are:

* Copanlisib
* Ibrutinib
* Acalabrutinib

DETAILED DESCRIPTION:
This is an open-label, phase II study, adding copanlisib to ibrutinib or acalabrutinib in select participants who are receiving ibrutinib for relapsed/refractory CLL.

Copanlisib has not been approved by the U.S. Food and Drug Administration (FDA) for CLL, but it has been approved for use in relapsed/refractory follicular lymphoma. Ibrutinib and acalabrutinib are approved by the FDA as a treatment option for CLL.

This research study is:

* Trying to understand what effects, good or bad, treatment with copanlisib in combination with ibrutinib or acalabrutinib has in select participants who are receiving ibrutinib for relapsed/refractory CLL
* Determining if this approach is better or worse than the usual approach for this type of cancer
* Determining whether genomic changes in CLL cells and changes in immune response make treatment with the study drugs more or less effective

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

Participants will receive combination therapy for six months before resuming ibrutinib alone. They will continue therapy for as long as they do not have serious side effects and their disease does not get worse and will be followed for up to 5 years.

It is expected that about 30 people will take part in this research study.

Bayer HealthCare Pharmaceuticals is supporting this research study by providing the study drug, copanlisib. Ibrutinib and acalabrutinib will be obtained from commercial supply.

ELIGIBILITY:
Inclusion Criteria:

* Must have a confirmed diagnosis of chronic lymphocytic leukemia or small lymphocytic lymphoma as per 2018 IWCLL criteria with evidence of persistent disease, defined as measurable adenopathy or splenomegaly, circulating disease, or marrow disease
* On ibrutinib or acalabrutinib which was instituted due to patient previously meeting 2018 IWCLL criteria for treatment, started at least 6 months prior to study entry for any patient who have received at least one prior line of therapy prior to ibrutinib or acalabrutinib. Reduced dose of ibrutinib or acalabrutinib is allowed as long as the dose has been stable for at least 4 weeks and all toxicities are ≤ grade 1
* Must have achieved either SD, PR or PR-L on ibrutinib or acalabrutinib by 2018 IWCLL criteria
* ECOG performance status < 2
* Patients must meet the following hematologic criteria at screening, unless they have significant bone marrow involvement of CLL confirmed on biopsy:

  * Absolute neutrophil count ≥500 cells/mm3 (0.5 x 109/L). Growth factor is allowed in order to achieve this
  * Platelet count ≥50,000 cells/mm3 independent of transfusion within 7 days of screening
* Adequate hepatic function defined as: Serum aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 x upper limit of normal (ULN), bilirubin ≤2.0 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin including hemolysis)
* Adequate renal function defined by serum creatinine ≤1.5 x ULN or creatinine clearance (by Cockroft-Gauldt ≥ 50 ml/min
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients receiving cancer therapy (i.e., chemotherapy, radiation therapy, immunotherapy, biologic therapy, hormonal therapy, surgery and/or tumor embolization) other than ibrutinib or acalabrutinib within 2 weeks of Cycle 1/Day 1 with the following exceptions:

  * Limited palliative radiation is allowed if completed > 1 weeks of C1D1
  * Hormonal therapy given in the adjuvant setting
  * Corticosteroid therapy (prednisone or equivalent <15 mg daily) is allowed as clinically warranted as long as the dose is stabilized at least for 7 days prior to initial dosing.Topical or inhaled corticosteroids are permitted
* Within six months of allogeneic hematologic stem cell transplant at the time of starting study treatment or active graft vs. host disease requiring systemic treatment or prophylaxis within 6 weeks of starting study treatment
* Prior treatment with copanlisib
* Patients in CR on ibrutinib or acalabrutinib
* History of other malignancies, except:

  * Malignancy treated with curative intent and with no known active disease present for ≥2 years before the first dose of study drug and felt to be at low risk for recurrence by treating physician
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease.
  * Low-risk prostate cancer on active surveillance
* Vaccinated with live, attenuated vaccines <4 weeks before first dose of study drug
* Active autoimmune disease requiring systemic treatment
* Recent infection requiring intravenous antibiotics that was completed ≤7 days before the first dose of study drug, or any uncontrolled active systemic infection
* Known bleeding disorders (eg, von Willebrand's disease) or hemophilia
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment
* Human immunodeficiency virus (HIV) or active hepatitis C virus (HCV) or hepatitis B virus (HBV) infection
* CMV PCR positive at baseline
* Major surgery within 4 weeks of first dose of study drug
* History of or concurrent condition of interstitial lung disease of any severity and/or severely impaired lung function (as judged by the investigator)
* Concurrent diagnosis of pheochromocytoma
* Uncontrolled arterial hypertension despite optimal medical management
* Type 1 or type 2 diabetes mellitus with a HgbA1c > 8.5%
* Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety
* Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to randomization
* Unable to swallow capsules or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction
* Lactating or pregnant
* Patients with known CNS involvement
* Concurrent administration of medications or foods that are strong inhibitors or inducers of CYP3A
* Known hypersensitivity to copanlisib, ibrutinib, or acalabrutinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) Rate | 6 months
  Rate of complete response (CR) by 2018 IWCLL criteria following the addition of six months of copanlisib to the therapy of patients with SD or PR or PR-L on ibrutinib or acalabrutinib in the relapsed/refractory setting.

SECONDARY OUTCOMES:
Number of Participants with Treatment Related Adverse Events as Assessed by CTCAE ver. 5.0. | 6 months
  Adverse events will be collected and reported as percentages
Duration of Response (DOR) | 3 years
  Legnth of time the patients respond to therapy
Progression-free Survival (PFS) | 3 years
  The time from registration to progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation.
Overall Survival (OS) | 3 years
  The time from registration to death due to any cause or censored at date last known alive.

CONTACTS AND LOCATIONS:
Overall Officials: Inhye Ahn, MD, Principal Investigator — Dana-Farber Cancer Institute

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu